CLINICAL TRIAL: NCT01670565
Title: Belimumab for the Treatment of Diffuse Cutaneous Systemic Sclerosis: A Phase 2a, Single-centered, Randomized, Placebo-controlled, Double-blind, Proof-of-concept Pilot Study.
Brief Title: Belimumab for the Treatment of Diffuse Cutaneous Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-279
Record Dates: First submitted 2012-08-15; First posted 2012-08-22 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Systemic Sclerosis
Keywords: Diffuse cutaneous systemic sclerosis; Early Diffuse cutaneous systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — belimumab; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate mofetil + Belimumab (Experimental): All patients who enroll in this trial will FIRST receive mycophenolate mofetil (MMF, Cellcept), which is a drug commonly given to patients with scleroderma in clinical practice. This drug will be given at no cost to the patient. After the patient has been titrated to 2 grams of MMF per day, the patient will receive EITHER a 10 mg/kg belimumab (Benlysta) intravenous infusion OR a placebo (saline) infusion. This medication and infusion will of course be covered by the study.
  Interventions: Drug: Belimumab; Drug: Mycophenolate Mofetil
- Mycophenolate Mofetil + Saline (placebo) (Placebo Comparator): In order to observe the difference between belimumab/MMF compared to MMF alone, half of the patients will receive a normal saline infusion that appears identical to the belimumab infusion.
  Interventions: Drug: Mycophenolate Mofetil; Other: Placebo Infusion

INTERVENTIONS:
Drug: Belimumab — Belimumab (Benlysta®) decreases B-Cell survival and has been FDA approved for the treatment of systemic lupus erythematosus, another rheumatic autoimmune disease. Belimumab is a recombinant, fully human monoclonal antibody; it binds to the soluble human B lymphocyte stimulator (BLyS) with high affinity and inhibits its biologic activity. Prior research provides a robust rationale for the investigation of belimumab in combination with MMF (Cellcept ®) for the treatment of early diffuse cutaneous systemic sclerosis.
  Other Names: Benlysta
  Arms: Mycophenolate mofetil + Belimumab
Drug: Mycophenolate Mofetil — Patients received background MMF therapy, some who were naive to MMF were titrated up to 1,000 mg twice daily and others had been receiving MMF at <2,000 mg/day for <3 months. MMF was chosen so that background therapy would be uniform and not a further source of variability in the small study.
  Other Names: MMF, Cellcept
Other: Placebo Infusion — Infusion of normal saline
  Arms: Mycophenolate Mofetil + Saline (placebo)

SUMMARY:
This is a 48 week, phase IIa, single center, randomized, double-blind, placebo-controlled, proof-of-concept pilot study. All participants will first be treated with mycophenolate mofetil (MMF, Cellcept) and titrated up to a dose of 2 grams/day. Following this period, half will be given either a belimumab (Benlysta®) or placebo intravenous infusion to treat early diffuse cutaneous systemic sclerosis. Belimumab/MMF is expected to improve disease activity measured by an improvement in skin thickening and stability of pulmonary function test measurements when compared to patients treated with placebo/MMF.

DETAILED DESCRIPTION:
The specific objectives of this study are to:

1. Determine whether belimumab used in combination with MMF is safe and tolerable in the treatment of patients with early diffuse cutaneous systemic sclerosis (Disease duration < 3 years).
2. Determine whether belimumab used in combination with MMF is more effective in the treatment of diffuse cutaneous systemic sclerosis than MMF alone, as measured by change in modified Rodnan Skin Score (mRSS), forced vital capacity (FVC), hemoglobin corrected diffusion capacity (DLCO), Medsger Severity Scale (MSS), and by other physician and patient derived outcome measures.
3. Determine the biological activity of Belimumab/MMF as assessed by effect on histology of skin, change in B-Cell profiles, effect on BLyS levels, and effect on serological and cutaneous biomarkers of disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to eighteen years.
2. Clinical diagnosis of diffuse systemic sclerosis by ACR criteria, with a stable modified Rodnan skin score in the one month preceding introduction of belimumab therapy.
3. Disease duration of less than or equal to 3 years as defined by the date of onset of the first non-Raynaud's symptom.

Exclusion Criteria:

1. Inability to render informed consent in accordance with institutional guidelines.
2. Disease duration of greater than 3 years.
3. Patients with mixed connective tissue disease or "overlap" (i.e. those who satisfy more than one set of ACR criteria for a rheumatic disease.)
4. Limited scleroderma.
5. Systemic sclerosis-like illness associated with environmental or ingested agents such as toxic rapeseed oil, vinyl chloride, or bleomycin.
6. Ongoing treatment with immunosuppressive therapies including cyclophosphamide, azathioprine, methotrexate, or cyclosporine, or use of those medications within 1 month of trial entry.
7. The use of other anti-fibrotic agents including colchicine, D-penicillamine, minocycline, tyrosine kinase inhibitors (nilotinib, imatinib, dasatinib), or Type 1 oral Collagen in the month prior to enrollment.
8. Use in the prior month of corticosteroids at doses exceeding the equivalent of prednisone 10 mg daily. Use of corticosteroid at < 10 mg of prednisone can continue during the course of the study.
9. Treatment with MMF at a dose of ≥ 2 grams daily for > 3 months.
10. Concurrent serious medical condition which in the opinion of the investigator makes the patient inappropriate for this study such as uncontrollable CHF, arrhythmia, severe pulmonary or systemic hypertension, severe GI involvement, hepatic impairment, serum creatinine of greater than 2.0, active infection, severe diabetes, unstable atherosclerotic cardiovascular disease, malignancy, HIV, or severe peripheral vascular disease.
11. A positive pregnancy test at entry into this study.
12. Men and women with reproductive potential will be required to use effective means of contraception through the course of the study, such as a tubal ligation or hysterectomy, condom or diaphragm used with a spermicide,or an intrauterine device (IUD). Approved hormonal contraceptives (such as birth control pills, patches, implants or injections) may interact with and reduce the effectiveness of MMF and thus, are not acceptable. Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use.
13. Breastfeeding. Breastfeeding is contraindicated with the use of MMF.
14. Participation in another clinical research study involving the evaluation of another investigational drug within ninety days of entry into this study.
15. The presence of severe lung disease as defined by a diffusion capacity of less than 30% of predicted or requiring supplemental oxygen.
16. History of HIV infection
17. Known active bacterial, viral, fungal, mycobacterial, or other infection r any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening, or oral antibiotics within 2 weeks prior to screening
18. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
19. Prior use of Belimumab, Rituximab, or other B-Cell depleting therapies ever
20. The use of other biologics including TNF inhibitors, abatacept, or tocilizumab within 1 month of enrollment [this is a safety issue]
21. Patients with a history of severe depression, psychosis, or suicidal ideation will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Spiera, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] Gordon JK, Martyanov V, Franks JM, Bernstein EJ, Szymonifka J, Magro C, Wildman HF, Wood TA, Whitfield ML, Spiera RF. Belimumab for the Treatment of Early Diffuse Systemic Sclerosis: Results of a Randomized, Double-Blind, Placebo-Controlled, Pilot Trial. Arthritis Rheumatol. 2018 Feb;70(2):308-316. doi: 10.1002/art.40358. Epub 2017 Dec 29. PMID 29073351
- See also: Scleroderma, Vasculitis, & Myositis Center Website — http://www.hss.edu/scleroderma-vasculitis-center.asp

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil + Belimumab: Patients in this arm will FIRST receive mycophenolate mofetil (MMF, Cellcept), which is a drug commonly given to patients with scleroderma in clinical practice titrated to 2 grams of MMF per day, followed by 10 mg/kg belimumab (Benlysta). Belimumab Infusion will be administered 14 times over a period of 48 weeks. MMF will be administered through 48 weeks.
  Belimumab: Belimumab (Benlysta®) decreases B-Cell survival and has been FDA approved for the treatment of systemic lupus erythematosus, another rheumatic autoimmune disease. Belimumab is a recombinant, fully human monoclonal antibody; it binds to the soluble human B lymphocyte stimulator (BLyS) with high affinity and inhibits its biologic activity. Prior research provides a robust rationale for the investigation of belimumab in combination with MMF (Cellcept ®) for the treatment of early diffuse cutaneous systemic sclerosis.
- Mycophenolate Mofetil + Saline (Placebo): Patients in this arm will FIRST receive MMF alone followed by normal saline infusion that appears identical to the belimumab infusion. Saline Infusion will be administered 14 times over a period of 48 weeks. MMF will be administered through 48 weeks.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo)
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Mycophenolate Mofetil + Belimumab: All patients who enroll in this trial will FIRST receive mycophenolate mofetil (MMF, Cellcept), which is a drug commonly given to patients with scleroderma in clinical practice. This drug will be given at no cost to the patient. After the patient has been titrated to 2 grams of MMF per day, the patient will receive EITHER a 10 mg/kg belimumab (Benlysta) intravenous infusion OR placebo (saline) infusion. This medication and infusion will be covered by the study.
  Belimumab: Belimumab (Benlysta®) decreases B-Cell survival and has been FDA approved for the treatment of systemic lupus erythematosus, another rheumatic autoimmune disease. Belimumab is a recombinant, fully human monoclonal antibody; it binds to the soluble human B lymphocyte stimulator (BLyS) with high affinity and inhibits its biologic activity. Prior research provides a robust rationale for the investigation of belimumab in combination with MMF (Cellcept ®) for the treatment of early diffuse cutaneous systemic sclerosis.
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12.1) | 56.7 (10.26) | 54.85 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20
Interstitial Lung Disease (ILD) [Count of Participants; unit: Participants] | 1 | 2 | 3
Anti-Scl-70 [Count of Participants; unit: Participants] — Characteristics of the patients at baseline. Number and percent of participants in each group who were positive for anti-Scl-70. The presence of anti-Scl-70 antibodies increases the risk for diffuse skin involvement and scleroderma related lung disease.
  Participants | 2 | 3 | 5
Anti- RNA Pol III [Count of Participants; unit: Participants] — Characteristics of the patients at baseline. Number and percent of participants in each group who were positive for Anti-RNA polymerase III. Numerous studies have shown that systemic sclerosis patients with anti-RNA polymerase III have an increased risk of the diffuse cutaneous form of scleroderma.
  Participants | 7 | 3 | 10
Modified Rodnan Skin Score (MRSS) at baseline [Median (Inter-Quartile Range); unit: units on a scale] — The Modified Rodnan Skin Score (MRSS) measures dermal skin thickness through the examination of 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (in pairs), and face, chest, and abdomen. The skin score is 0 for uninvolved skin through 3 for severe thickening (hidebound skin). The total skin score is the sum of the skin scores of the individual areas. The minimum score is 0 and the maximum score is 51. A higher score indicates greater severity of disease. Population: MRSS values are given for treated patients (n=9 per group) and not for all patients randomized (n=10 per group)
  units on a scale
    number analyzed (Participants) | 9 | 9 | 18
    (all) | 27 [26.5 to 31] | 28 [22 to 28] | 27 [22 to 29]
Forced Vital Capacity (FVC) [Median (Inter-Quartile Range); unit: % predicted] — FVC % predicted at baseline. Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from the lungs after taking a deep breath. It is used to determine the severity of lung disease. FVC for a given individual is compared to reference or predicted values. The reference values are based on healthy individuals with normal lung function and indicates values that would be expected for someone of the same sex, age and height. FVC % predicted compares the patients FVC values with the reference values. Population: Values for treated patients such as FVC% predicted and DLCO% predicted are given for treated patients (n=9 per group) and not for all patients randomized (n=10).
  % predicted
    number analyzed (Participants) | 9 | 9 | 18
    (all) | 88 [81 to 100] | 95 [88 to 101] | 94.5 [81 to 101]
Diffusing capacity of the lungs for carbon monoxide [Median (Inter-Quartile Range); unit: % predicted] — Diffusing capacity of the lungs for carbon monoxide (DLCO) measures how much oxygen travels from the alveoli of the lungs to the blood stream. It is used to determine the severity of lung disease. DLCO for a given individual is compared to reference values. The reference values are based on healthy individuals with normal lung function and indicates values that would be expected for someone of the same sex, age and height. DLCO % predicted compares the patients DLCO values with the reference values. An individuals DLCO result that is at least 80% of the predicted value is considered normal. Population: Values for treated patients such as FVC% predicted and DLCO% predicted are given for treated patients (n=9 per group) and not for all patients randomized (n=10).
  % predicted
    number analyzed (Participants) | 9 | 9 | 18
    (all) | 85 [67 to 94] | 81 [81 to 87] | 83 [67 to 92]

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Rodnan Skin Score (MRSS)
Description: Change in MRSS is measured by median change (and interquartile range) from Baseline median to week 52 median. The efficacy of the drug will be measured as the change in the Modified Rodnan Skin Score (MRSS) at 52 weeks. The Modified Rodnan Skin Score (MRSS) measures dermal skin thickness through the examination of 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (in pairs), and face, chest, and abdomen. The skin score is 0 for uninvolved skin through 3 for severe thickening (hidebound skin). The total skin score is the sum of the skin scores of the individual areas. The minimum score is 0 and the maximum score is 51. A higher score indicates greater severity of disease
Time Frame: Baseline and at 52 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Mycophenolate Mofetil + Belimumab: All patients who enroll in this trial will FIRST receive mycophenolate mofetil (MMF, Cellcept), which is a drug commonly given to patients with scleroderma in clinical practice. This drug will be given at no cost to the patient. After being titrated to 2 grams of MMF per day, patients in this experimental group will receive a 10 mg/kg belimumab (Benlysta) intravenous infusion infusion.This medication and infusion will of course be covered by the study.
  Belimumab: Belimumab (Benlysta®) decreases B-Cell survival and has been FDA approved for the treatment of systemic lupus erythematosus, another rheumatic autoimmune disease. Belimumab is a recombinant, fully human monoclonal antibody; it binds to the soluble human B lymphocyte stimulator (BLyS) with high affinity and inhibits its biologic activity. Prior research provides a robust rationale for the investigation of belimumab in combination with MMF (Cellcept ®) for the treatment of early diffuse cutaneous systemic
- Mycophenolate Mofetil + Saline (Placebo): In order to observe the difference between belimumab/MMF compared to MMF alone, half of the patients will receive a normal saline infusion that appears identical to the belimumab infusion.
  All patients who enroll in this trial will FIRST receive mycophenolate mofetil (MMF, Cellcept), which is a drug commonly given to patients with scleroderma in clinical practice. This drug will be given at no cost to the patient. After being titrated to 2 grams of MMF per day, patients in this experimental group will receive a placebo (saline) infusion.This infusion will of course be covered by the study.
  .
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo)
Number analyzed (Participants) | 10 | 10
units on a scale | -10 [-13 to -9] | -3.0 [-15 to -1]

2. Primary Outcome: Number of Adverse Events and Serious Adverse Events
Description: The safety and tolerability of belimumab in patients with systemic sclerosis will be as assessed by comparing the rates of adverse events (AEs) and serious adverse events (SAEs) between treatment and placebo groups.
Time Frame: At 52 weeks
Measure: Number; unit: number of AEs
Groups:
- Mycophenolate Mofetil + Saline (Placebo): In order to observe the difference between belimumab/MMF compared to MMF alone, half of the patients will receive a normal saline infusion that appears identical to the belimumab infusion.
  All patients who enroll in this trial will FIRST receive mycophenolate mofetil (MMF, Cellcept), which is a drug commonly given to patients with scleroderma in clinical practice. This drug will be given at no cost to the patient. After being titrated to 2 grams of MMF per day, patients in this experimental group will receive a placebo (saline) infusion.This infusion will of course be covered by the study.
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo)
Number analyzed (Participants) | 10 | 10
number of AEs
  Total number of AEs | 53 | 56
  Total number of infectious AEs | 18 | 16
  Serious AEs | 0 | 3

3. Primary Outcome: Change in Forced Vital Capacity (FVC)
Description: Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from the lungs after taking a deep breath. It is used to determine the severity of lung disease. FVC for a given individual is compared to reference or predicted values. The reference values are based on healthy individuals with normal lung function and indicates values that would be expected for someone of the same sex, age and height. FVC % predicted compares the patients FVC values with the reference values. Results are considered normal if FVC is 80 percent or more of the predicted value. Change in FVC % predicted is measured by median change (and interquartile range) from Baseline median to week 52 median.
Time Frame: Baseline and Week 52
Measure: Median (Inter-Quartile Range); unit: % predicted
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo)
Number analyzed (Participants) | 9 | 9
% predicted | 5.00 [0.00 to 8.00] | -2.00 [-6.00 to 4.00]

4. Primary Outcome: Change in Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO)
Description: Diffusing capacity of the lungs for carbon monoxide (DLCO) measures how much oxygen travels from the alveoli of the lungs to the blood stream. It is used to determine the severity of lung disease. DLCO for a given individual is compared to reference or predicted values. The reference values are based on healthy individuals with normal lung function and indicates values that would be expected for someone of the same sex, age and height. DLCO % predicted compares the patients DLCO values with the reference values. An individuals DLCO result that is at least 80% of the predicted value is considered normal. Change in DLCO % predicted is measured by median change (and interquartile range) from Baseline median to week 52 median.
Time Frame: Baseline and Week 52
Measure: Median (Inter-Quartile Range); unit: % predicted
Groups:
- Mycophenolate Mofetil + Belimumab: All patients who enroll in this trial will FIRST receive mycophenolate mofetil (MMF, Cellcept), which is a drug commonly given to patients with scleroderma in clinical practice. This drug will be given at no cost to the patient. After being titrated to 2 grams of MMF per day, the patient will receive a 10 mg/kg belimumab (Benlysta) intravenous infusion.This medication and infusion will of course be covered by the study.
  Belimumab: Belimumab (Benlysta®) decreases B-Cell survival and has been FDA approved for the treatment of systemic lupus erythematosus, another rheumatic autoimmune disease. Belimumab is a recombinant, fully human monoclonal antibody; it binds to the soluble human B lymphocyte stimulator (BLyS) with high affinity and inhibits its biologic activity. Prior research provides a robust rationale for the investigation of belimumab in combination with MMF (Cellcept ®) for the treatment of early diffuse cutaneous systemic
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo)
Number analyzed (Participants) | 9 | 9
% predicted | 2.00 [-7.00 to 7.00] | 0.00 [-6.00 to 7.00]

5. Secondary Outcome: Change in Scleroderma Health Assessment Questionnaire Disability Index (SHAQ DI)
Description: The Scleroderma Health Assessment Questionnaire (SHAQ) consist of the Health Assessment Questionnaire (HAQ) and 8 other domains addressing scleroderma related manifestations that contribute to disability. It is a quality of life measure. Each question is scored from 0 (without difficulty) to 3 (unable to do). Some domains in the SHAQ are visual analog scales that are measured first and then changed to a 0-3 scale.
  The maximum from each category is added together and divided by the number of categories completed. The total scale range is 0-3. A higher score indicates worse functionality.
  Change in Scleroderma Health Assessment Questionnaire Disability Index (SHAQ-DI) is measured as median change (and interquartile range) from Baseline median to week 52 median. The reported median change can range from -3 to 3. A negative median change indicates a better outcome.
Time Frame: Baseline and Week 52
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo)
Number analyzed (Participants) | 9 | 9
score on a scale | -0.25 [-0.38 to -0.25] | 0.00 [-0.13 to 0.13]

6. Secondary Outcome: Change in in Short Form-36 (SF-36) Questionnaire:Mental Component Summary
Description: The Short Form 36 (SF-36) is a validated 36 item questionnaire which measures quality of life across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health. The mental component score (MCS) is composed of a subset of the 8 health domains. Each component is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 is equivalent to no disability. The SF-36 mental component can be obtained by looking at the mean average of all the emotionally relevant items. Change in Short Form 36 mental (SF-36 MC) is measured by median change (and interquartile range) from Baseline to week 52. The median change can range from -100 to 100. A positive median change indicates indicates an improved outcome.
Time Frame: Baseline and at 52 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo)
Number analyzed (Participants) | 9 | 9
score on a scale | 7.50 [2.50 to 18.50] | 3.00 [0.00 to 10.00]

7. Secondary Outcome: Change in Short Form-36 (SF-36) Questionnaire: Physical Component Summary
Description: The Short Form 36 (SF-36) is a 36 item questionnaire which measures quality of life across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health. The physical component score is composed of a subset of the 8 health domains.The SF-36 physical component can be obtained by looking at the mean average of all the physically relevant items. Each component is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 is equivalent to no disability. Change in Short Form 36 physical component (SF-36 PC) is measured by median change (and interquartile range) from Baseline to week 52. The median change can range from -100 to 100. A positive median change indicates indicates an improved outcome.
Time Frame: Baseline and Week 52
Measure: Median (Inter-Quartile Range); unit: scores on a scale, 0-100
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo)
Number analyzed (Participants) | 9 | 9
scores on a scale, 0-100 | 8.00 [-3.50 to 19.00] | -3.00 [-3.00 to 27.00]

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Mycophenolate Mofetil + Belimumab: All patients who enroll in this trial will FIRST receive mycophenolate mofetil (MMF, Cellcept), which is a drug commonly given to patients with scleroderma in clinical practice. This drug will be given at no cost to the patient. After being titrated to 2 grams of MMF per day, the patient will receive a 10 mg/kg belimumab (Benlysta) intravenous infusion. This medication and infusion will be covered by the study.
  Belimumab: Belimumab (Benlysta®) decreases B-Cell survival and has been FDA approved for the treatment of systemic lupus erythematosus, another rheumatic autoimmune disease. Belimumab is a recombinant, fully human monoclonal antibody; it binds to the soluble human B lymphocyte stimulator (BLyS) with high affinity and inhibits its biologic activity. Prior research provides a robust rationale for the investigation of belimumab in combination with MMF (Cellcept ®) for the treatment of early diffuse cutaneous systemic sclerosis.
Arm/Group | Mycophenolate Mofetil + Belimumab | Mycophenolate Mofetil + Saline (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/10
Other Adverse Events (participants affected / at risk) | 9/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil + Belimumab (N=10) | Mycophenolate Mofetil + Saline (Placebo) (N=10)
Anxiety Attack (Psychiatric disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) — related to progression of SSc-related cardiomyopathy
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — related to progression of SSc-related cardiomyopathy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil + Belimumab (N=10) | Mycophenolate Mofetil + Saline (Placebo) (N=10)
Urinary Tract Infection (Renal and urinary disorders) | 2 (3) | 3 (6)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Vomiting (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (3)
Nausea (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Zoster (Infections and infestations) | 1 (1) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Lymphocyte count decreased (Immune system disorders) | 1 (1) | 2 (2)
Lip infection (HSV-1) (Infections and infestations) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Allergic Reaction (Infusion) (General disorders) | 1 (1) | 0 (0)
ALT Increased (General disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
AST Increased (General disorders) | 1 (1) | 0 (0)
Asymptomatic Bacteriuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Conjunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Gastroesophageal Refluex Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemoglobin A1c Increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IgM Decreased (Immune system disorders) | 1 (1) | 0 (0)
Infections and Infestations -Other (H Pylori, Stomach) (Infections and infestations) | 1 (1) | 0 (0)
Infections and Infestations -Other (Viral Syndrome) (Infections and infestations) | 1 (1) | 0 (0)
Laryngeal Inflammation (Infections and infestations) | 1 (1) | 0 (0)
Meniscal Tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acroosteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Calcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oral Hemorrhage (General disorders) | 1 (1) | 0 (0)
Otitis Media (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pulmonary Nodule Benign (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Salivary Gland Infection (Infections and infestations) | 1 (1) | 0 (0)
Testicular Disorder (hydrocele) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Tooth Mobility (General disorders) | 1 (1) | 0 (0)
Anxiety (Acute) (Psychiatric disorders) | 0 (0) | 1 (1)
Aortic Valve Disease (progression) (Vascular disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Chest-Pain Cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CPK Increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fracture (Shoulder) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hermaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Irregular Menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Irritable Bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Memory Impairment-acute (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Skin Ulceration (Leg) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Soft Tissue Infection (wart) (Infections and infestations) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (General disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Vaginal Infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Weight Loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes